CLINICAL TRIAL: NCT04396184
Title: Conventional Photodynamic Therapy vs. Painless Photodynamic Therapy for Actinic Keratosis#a Randomized, Open-label Trial
Brief Title: Conventional Photodynamic Therapy vs. Painless Photodynamic Therapy for Actinic Keratosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Dermatology Hospital (Other)
Responsible Party: Principal Investigator, Xiuli Wang, Director, Clinical Professor, Shanghai Dermatology Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020-09
Record Dates: First submitted 2020-05-17; First posted 2020-05-20 (Actual); Last update posted 2020-05-20 (Actual); Status verified 2020-05

CONDITIONS: Actinic Keratosis
Keywords: Photodynamic Therapy; Conventional; Painless; Actinic Keratosis
MeSH Terms: conditions — Keratosis, Actinic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Evaluator assesses photographs without prior knowledge of intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Painless Photodynamic Therapy(P-PDT) group (Experimental): The painless photodynamic therapy group underwent narrow-band light-emitting diode (LED) irradiation (630 nm; 288 J/cm2) after applying 5% 5-aminolevulinic acid#ALA#cream for 30min. A repeat treatment was administered once every two weeks for 3 times.
  Interventions: Procedure: Aminolevulinic acid photodynamic therapy
- Conventional Photodynamic Therapy(C-PDT) group (Active Comparator): The conventional photodynamic therapy(C-PDT) group underwent narrow-band light-emitting diode (LED) irradiation (630 nm; 140 J/cm2) after applying 5% 5-aminolevulinic acid cream for 3h.A repeat treatment was administered once every two weeks for 3 times.
  Interventions: Procedure: Aminolevulinic acid photodynamic therapy

INTERVENTIONS:
Procedure: Aminolevulinic acid photodynamic therapy — Aminolevulinic acid photodynamic therapy

SUMMARY:
This study is being done to compare a new, continuous illumination and short Incubation time regimen of aminolevulinic acid photodynamic therapy#ALA-PDT) to a conventional regimen for treatment of Actinic Keratosis. The hypothesis is that the continuous illumination approach will be less or even no painful, but equally efficacious, as the old regimen.

DETAILED DESCRIPTION:
This study is being done to compare a new, continuous illumination and short Incubation time regimen of aminolevulinic acid photodynamic therapy#painless-PDT) to a conventional regimen for treatment of Actinic Keratosis. The hypothesis is that the continuous illumination approach will be less or even no painful, but equally efficacious, as the old regimen.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosed with AK (OLSEN classification grade I, II, III), aged > 18 years (Because no dosing or adverse event data are currently available on the use of topical aminolevulinic acid in patients <18 years of age, children are excluded from this study);
2. All patients are unfit and reluctant to undergo surgery for any reasons, and volunteered to participate in the study and ability to understand and the willingness to sign a written informed consent. Patents are willing to pay for the treatment, and agreed to take a picture of the skin lesions.

Exclusion Criteria:

1. Those who had ALA-PDT and any other studies that affect this study within 12 weeks ;
2. There are other facial diseases that may affect the efficacy evaluation, such as other photodermatosis;
3. Take phototoxic or photosensitizer within 8 weeks;
4. Clinical and / or pathological prove that the tumor has invaded other organs or tissues;
5. Serious immunocompromised persons;
6. scar constitution;
7. Patients are known to have skin photosensitivity, porphyria, or allergies to ALA, light or lidocaine;
8. Persons are suffering from severe internal diseases, mental and mental illness, infectious diseases or pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2020-05-01 (Actual); Primary Completion 2021-04-30 (Estimated); Study Completion 2021-04-30 (Estimated)

PRIMARY OUTCOMES:
The clearance rate of Actinic Keratoses | six weeks after treatment
  The change rate in lesion clearance of Actinic Keratoses at six weeks after treatment will be measured as the primary outcome

SECONDARY OUTCOMES:
Pain assessment | Immediately, 1st minute, 3rd minute, 5th minute, 10th minute, 30th minute, 1hour ,2hour, 4hour, 12hour, 24hour,48hour ,72hour
  The pain will be assessed using Vissual Analogue Scale(VAS) with a score range of 0-10.The higher the score,the greater the pain, with 0 being no pain and 10 being the most unbearable pain. Pain will be measured at different time points during and after every treatment

CONTACTS AND LOCATIONS:
Overall Officials: Xiuli Wang, PHD,MD, Study Chair — Shanghai Skin Disease Hospital
Locations (1):
- Yunfeng Zhang, Shanghai, Jinan, China

IPD SHARING:
Plan to Share IPD: Yes
underlie results
Supporting Information: CSR
Time Frame: One year after finishing this srudy and for permanency
Access Criteria: anyone who search pubmed